CLINICAL TRIAL: NCT02266251
Title: Optimizing Health Outcomes in Patients With Symptomatic Aortic Valve Disease
Acronym: PCORI-AVR
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); American College of Cardiology (Other); The Society of Thoracic Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00052757; CER-1306-04350 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-10-13; First posted 2014-10-16 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical AVR: No interventions will be administered. Retrospective data analysis will be completed to compare health outcomes among patients with a similar baseline health satus who are eligible for both procedures (operative transcatheter AVR patients enrolled in the Transcatheter Valve Therapies (TVT) Registry (Nov 2011-Dec 2013) and surgical AVR patients with STS perioperative risk of mortality whose index procedure is included in the STS Adult Cardiac Surgical DAtabase (ACSD) (Jan 2011-Dec 2013).
- Transcatheter AVR: No interventions will be administered. Retrospective data analysis will be completed to compare health outcomes among patients with a similar baseline health satus who are eligible for both procedures (operative transcatheter AVR patients enrolled in the TVT Registry (Nov 2011-Dec 2013) and surgical AVR patients with STS perioperative risk of mortality whose index procedure is included in the STS ACSD (Jan 2011-Dec 2013).

SUMMARY:
Disease of the aortic heart valve is both common and progressively disabling, with no effective medical treatment. In November 2011, the United States Food and Drug Administration (U.S. FDA) approved a new, less invasive transcatheter alternative to surgical aortic valve replacement (AVR). This new technology has changed the treatment of patients with aortic valve disease. In doing so, it has created a pressing clinical need for shared decision making tools that will help patients understand the risks and benefits of each treatment alternative in the setting of their individual characteristics.

The overarching goal of this study is to develop a new way to approach the treatment of medical illness, by focusing on the expected treatment outcomes for individual patients using information collected from large groups of patients. The corner-stone of this model is a public website that is designed to engage patients and clinicians in a personalized discussion of treatment alternatives. To achieve this goal for patients with aortic valve disease, we will use existing clinical data from the Society of Thoracic Surgeons (STS) and American College of Cardiology (ACC) national procedural registries that has been linked to Medicare claims for patient follow-up to 1) evaluate important health outcomes with surgical versus transcatheter AVR among patients who would be eligible for surgical AVR, and 2) create and evaluate personalized decision assistance tools for all patients considering AVR. This work will be accomplished in direct partnership with both patients and caregivers as well as a diverse group of stakeholders who will help ensure its usefulness and dissemination.

DETAILED DESCRIPTION:
Aortic valve disease is a common, progressively debilitating condition with no effective medical treatment. Surgical aortic valve replacement (AVR) has been the standard of care in the presence of valve-associated symptoms which include heart failure, chest pain, and syncope; however, in November 2011, long-standing treatment algorithms were disrupted with the United States Food and Drug Administration (U.S. FDA) approval of a less invasive transcatheter alternative to surgical aortic valve replacement (AVR) with a different profile of associated risks and benefits. This new technology has created a pressing clinical need for shared decision making tools to help translate the "average-patient" clinical trial results to more relevant "patient-specific" information that will empower individuals facing this important treatment decision.

The overarching goal of this study is to develop a broadly applicable patient-centered paradigm for the treatment of medical illness. The corner-stone of this model is an open-access, web-based resource to engage patients, their caregivers, and clinicians in a personalized treatment discussion. To achieve this goal for patients with aortic valve disease, we will use existing Medicare-linked clinical data from the Society of Thoracic Surgeons (STS) and American College of Cardiology (ACC) national procedural registries. This work will be accomplished in direct collaboration with patient and caregiver coinvestigators and a diverse stakeholder panel to ensure wide utility and dissemination.

Specifically, we will achieve the following three research aims:

Specific Aim 1. Compare contemporary health outcomes with surgical versus transcatheter AVR among operable patients in the United States; Specific Aim 2. Create and assess a personalized decision assistance tool to evaluate expected health outcomes with surgical vs. transcatheter AVR for operable patients with aortic valve disease; Specific Aim 3.Develop and assess a personalized risk assessment tool to evaluate expected health outcomes with transcatheter AVR for inoperable patients with aortic valve disease.

Additionally, we will achieve the general objective to create and evaluate web- and print-based educational resources for targeted dissemination to patients with aortic stenosis, their caregivers, and their healthcare providers.

The proposed research will facilitate a better match of patients with existing treatments and empower patients to actively participate in their own healthcare decisions, thereby improving the care of patients with aortic valve disease and reducing overall healthcare expenditures. This study will serve as a model to promote personalized medicine among both cardiovascular and non-cardiovascular disease states.

This study involves three primary comparisons. The first is a treatment comparison of surgical vs. transcatheter AVR on short and intermediate-term outcomes (stratified across important population subgroups)-important because the results will inform treatment discussions and decisions in vulnerable patients. The second is a comparison of outcomes across comorbidity sets using risk models-important because the resulting decision assistance tools will provide personalized estimates of risk to patients, caregivers, and providers as they select a treatment strategy. The third is an impact evaluation of an educational resource, including comparison of the change in treatment selection patterns and clinical outcomes across hospitals and geographic regions with high vs. low use of a web based educational resource-important because the comparison will provide critical pilot information to evaluate and tailor the resource impact.

ELIGIBILITY:
Inclusion Criteria:

* 'operable' transcatheter AVR patients enrolled in the TVT Registry (Nov 2011 -Dec 2013)
* surgical AVR patients with a STS perioperative risk of mortality (PROM) ≥4% whose index procedure is included in the STS ACSD (Jan 2011 - Dec 2013)

Exclusion Criteria:

* We will exclude patients with endocarditis or emergency/salvage status because these patients are rarely treated using transcatheter AVR in the United States (<0.2% incidence of either condition during the first year of TVT Registry data).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: To compare health outcomes among patients with a similar baseline health status who are eligible for surgical and transcather AVR procedures, we will include 1)'operable' transcatheter AVR patients enrolled in the TVT Registry (Nov 2011 -Dec 2013), and 2) surgical AVR patients with a STS perioperative risk of mortality (PROM) ≥4% whose index procedure is included in the STS ACSD (Jan 2011 - Dec 2013).
Sampling Method: Non-Probability Sample
Enrollment: 273365 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Mortality | one-year survival
  All-cause mortality will be analyzed in a time-to event analysis. Mortality follow-up will be considered to be administratively censored on the last date of Medicare follow-up which is expected to be 12/31/2013 for both surgical and transcatheter AVR.

SECONDARY OUTCOMES:
Stroke | during 1st year after surgical or transcatheter AVR
  incidence of a clinically apparent stroke
Discharged to home following the procedure (TAVR or SAVR) | STS ACSD (July 2011-June 2012) and STS/ACC TVT Registry (Nov 2011-March 2013)
  The percentage of patients discharged to home after TAVR versus SAVR will be estimated.
days alive and out of the hospital during the first post-operative year | number of days (out of 365) that the patient is alive and out of hospital during the first year post-operatively
  Among patients who were admitted from home, number of days (out of 365) that patient is alive and out of hospital during the first year post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: James M Brennan, MD, MPH, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No